CLINICAL TRIAL: NCT06757114
Title: A Study on the Multi-omic Factors Influencing the Efficacy of Immunotherapy and Adverse Reactions of Immunotherapy in Patients with Primary Non-small Cell Lung Cancer in High-altitude Areas
Brief Title: A Study on the Efficacy of Immunotherapy, the Occurrence and Severity of Adverse Reactions in Patients with Non-small Cell Lung Cancer in High-altitude Areas
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: （2024）EC-KY（NO.076）
Record Dates: First submitted 2024-12-10; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: High altitude — High altitude is defined as a long-term residence with an altitude of 1500m and above

SUMMARY:
As a major disease with high incidence and mortality rate, lung cancer seriously threatens the health of our people and causes a huge burden of disease. In recent years, with the widespread use of immune checkpoint inhibitors (ICIs), great progress has been made in the treatment of lung cancer, which has brought significant survival benefits to patients. Although ICI has greatly improved the prognosis of lung cancer patients, due to the complexity of the mechanism of action of ICI and the heterogeneity within the tumor, the benefit population of treatment is relatively limited, and some patients are still at risk of primary drug resistance and tumor hyperprogression.In this study, we aimed to compare the differences in the efficacy and adverse reactions of immunotherapy in patients with advanced non-small cell lung cancer at high and low altitudes, and to find out the relevant factors from multiple omics such as imaging, pathology, and genetics, so as to solve the problem of immunotherapy resistance

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with primary non-small cell lung cancer (adenocarcinoma/squamous cell carcinoma/adenosquamous cell carcinoma/large cell lung cancer/others) with clear cellular/histopathological evidence; (2) Primary non-small cell lung cancer of any stage receiving immunotherapy for the first time; (3) Patients who have undergone at least 2 cycles of immunotherapy during the treatment period and have undergone one efficacy evaluation; (4) Patients with at least one evaluable target lesion (except for those with uncontrolled brain metastases) according to Response Evaluation Criteria for Solid T Tumors (RECIST, version 1.1); (5) Voluntary participation in research and strong willingness to cooperate; (6) has been residing in Qinghai Province since birth; (7) Have been residing in Shaanxi Province since birth; (8) Be at least 18 years old;

Exclusion Criteria:

1. Patients with unknown histopathological type were excluded;
2. Patients with unclear diagnosis and treatment information and immunotherapy-related adverse reactions;
3. Patients with bipolar/multiple primary non-small cell lung cancer with other tumors were excluded;
4. Patients who are unwilling to join the study and have poor willingness to cooperate;
5. Patients who migrated to Qinghai or Shaanxi from different altitudes and had a history of migration between the two provinces were excluded;
6. exclude patients with a history of emigration from parents;
7. Patients who have received immunotherapy for other tumors in the past;
8. Prior immunosuppressive therapy prior to exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer receiving first-line immunotherapy at high and low altitudes
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of first-line immunotherapy for advanced non-small cell lung cancer at high and low altitudes | 2024/10/1-2025/3/31:Data Collection；2025/4/1-2025/6/3:Preliminary analysis；
  The evaluation indicators included progression-free survival(PFS), overall survival(OS), objective response rate(ORR), and disease conrtol rate(DCR)

SECONDARY OUTCOMES:
Immune-related adverse reactions in patients with non-small cell lung cancer receiving first-line immunotherapy at high and low altitudes | 2024/10/1-2025/3/31:Data Collection；2025/4/1-2025/6/3:Preliminary analysis；
  Type and severity of immune-related adverse effects

IPD SHARING:
Plan to Share IPD: No